CLINICAL TRIAL: NCT01660347
Title: Compassionate Use of the CliniMACS® CD34 Reagent System for Patients Requiring a Post Hematopoietic Stem Cell Transplant Boost of Donor Hematopoietic Stem Cells
Brief Title: Donor Stem Cell Boost in Treating Patients With Low Blood Cells After Donor Stem Cell Transplant
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 12D.214; 2012-35 (Other: CCRRC); JT 2962 (Other: JeffTrial Number)
Record Dates: First submitted 2012-08-05; First posted 2012-08-08 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Anemia; Hematopoietic/Lymphoid Cancer; Lymphopenia; Neutropenia; Thrombocytopenia
MeSH Terms: conditions — Anemia; Hematologic Neoplasms; Lymphopenia; Neutropenia; Thrombocytopenia | interventions — Peripheral Blood Stem Cell Transplantation; Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (allogeneic PBSCT boost) (Experimental): Patients undergo allogeneic PBSCT boost from cells selected for CD34+ using the CliniMACS CD34 Reagent System.
  Interventions: Biological: Allogeneic hematopoietic stem cell transplantation; Biological: Peripheral blood stem cell transplantation; Procedure: Management of therapy complications

INTERVENTIONS:
Biological: Allogeneic hematopoietic stem cell transplantation — Undergo allogeneic PBSCT boost using the CliniMACS CD34 Reagent System
Biological: Peripheral blood stem cell transplantation — Undergo allogeneic PBSCT boost using the CliniMACS CD34 Reagent System
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation; peripheral blood stem cell
Procedure: Management of therapy complications — Undergo allogeneic PBSCT boost using the CliniMACS CD34 Reagent System

SUMMARY:
This clinical trial studies how well donor stem cell boost works in treating patients with low blood cells after donor stem cell transplant. Donor stem cell boost may increase low blood cell counts caused by hematologic cancer or its treatment.

DETAILED DESCRIPTION:
Successful engraftment after allogeneic hematopoietic stem cell transplant (HSCT) is defined by an actual neutrophil count (ANC) of > 500 10^6/L and a self-sustaining platelet count of 20 x 10^9/L. ANC recovery usually occurs 14 to 21 days after the infusion of donor HSCs with red cell and platelet recovery typically following within the same time frame, although resolution of anemia may occur last. Recovery time is dose dependent, but in one report, donor HSC aliquots containing 1.9 to 20.5 10^6/kg CD34+ cells resulted in an ANC of > 500 10^6/L at a median of 12 days and 16 days for patients receiving filgrastim versus those not receiving a white cell growth factor. In this trial, self-sustaining platelet counts of 20 x 10^9/L occurred at median times of 15 to 11 days respectively. The results of another trial comparing outcomes between patients receiving mobilized peripheral blood stem cells (PBSCs) versus those receiving marrow from their donors showed that median times ANC of > 500 10^6/L and self-sustaining platelet counts of 20 x 10^9/L were 16 and 13 days respectively in the group receiving PBSCs and 21 and 19 days in those receiving marrow. Similar HSC doses associated with successful engraftment in these time frames have been demonstrated in other trials.

Most transplant centers require a minimum dose of 1 to 2 x 10^6 CD34+ cells/kg to achieve adequate count recovery in a reasonable time frame post HSCT, although an early trial examining recovery after autologous reinfusion of HSCs demonstrated that a threshold of 2.5 x 10^6/kg of CD 34 cells was associated with consistent and rapid WBC and platelet recovery times (18 and 14 days respectively). A later trial assessing autologous PBSC mobilization in breast cancer patients showed that HSC doses of ≥ 5 x 10^6 CD34+ cells/kg were associated with an 85% probability of WBC and platelet recovery by day 14, but with doses of 2 x 10^6 or less, 10% of patients had platelet recovery beyond day +28. While the precise dose of HSCs for successful engraftment in the allogeneic setting is not known, patient characteristics such as myelofibrosis and/or splenomegaly are likely to cause interpatient variation in the minimum number of HSCs needed for successful engraftment. In addition, donor factors such as mismatch in size with the recipient and biologic variation in the number of HSCs that can be obtained from any individual donor, can create a deficit in the amount of HSCs required for robust count recovery in a particular recipient. All of these factors can contribute to a poor functional or numeric cell dose and result in pancytopenia after HSCT.

Drugs required for the prophylaxis and treatment of GVHD and infection have myelotoxic effects post HSCT, and unlike their use in solid organ transplantation, the marrow toxic effects of these drugs are potentially more severe and longer lasting in the presence of a newly reconstituting immune system. While many drugs can have negative effects on marrow function after HSCT, mycophenolate mofetil (MMF) and ganciclovir are two of the most commonly used agents with the potential to cause cytopenias.

After hydrolysis to its active form, mycophenolic acid (MPA), MMF inhibits T and B cell proliferation making its use valuable in the prevention of graft versus host and host versus graft reactions post HSCT, especially in conjunction with a calcineurin inhibitor. Levels of MPA are increased in the presence of altered renal function, and other commonly used post HSCT drugs including acyclovir, ganciclovir, valaganciclovir, and tacrolimus. A major side effect of MMF is pancytopenia, particularly neutropenia, which is exacerbated by high drug levels. Due to finding of a wide interpatient variability in drug exposure, it has recently been recommended that the monitoring of MPA levels would result in better therapeutic outcomes, although MPA drug levels are not commonly obtained as yet in clinical practice. Myelotoxicity from the drug is observed after renal transplantation in the presence of a non-transplanted immune system demonstrating the potent myelosuppression associated with this drug, and the increased toxicity in patients with abnormal renal function. Patients post HSCT are treated with multiple drugs that both increase MPA levels and alter creatinine clearance, and are thereby highly susceptible to the marrow toxic effects of the drug which can result in cytopenias.

Ganciclovir and valganciclovir, which is rapidly converted to ganciclovir by intestinal mucosal cells and hepatocytes to ganciclovir, are inhibitors of DNA synthesis. Ganciclovir is a known myelotoxic drug that is effective in prophylaxis and treatment of cytomegalovirus (CMV) infections in transplant recipients. Salzberger et al. examined the outcomes between engraftment and day +100 post HSCT of 278 patients receiving ganciclovir and found that 41% of patients receiving the drug had an ANC less than 1000 10^6/L for at least 2 consecutive days. Hyperbilirubinemia during the first 20 days after HSCT, elevated serum creatinine after day +21, and low marrow cellularity between days +21 and +28 were significant risk factors for neutropenia. Patients with 3 risk factors had a 57% chance of developing neutropenia, which was significantly associated with a decreased overall and event free survival. As noted above, concomitant use of ganciclovir and MMF increase the serum concentration of both drugs exacerbating marrow toxicity. Because CMV is a life-threatening disease post HSCT, it is often necessary to use ganciclovir especially in the presence of renal failure which is exacerbated with the use of foscarnet, the alternate drug for CMV treatment. Therefore, ganciclovir-induced pancytopenia may be unavoidable in certain contexts.

Other medications with potentially toxic effects on the marrow alone or in combination with other commonly used agents which may contribute to the development of post HSCT cytopenias include levetiracetam, methotrexate, antibiotics such as linezolid, vancomycin, amoxicillin, cephalosporins, cidofovir, and gabapentin.

In addition to insufficient allogeneic cell doses and medication toxicities, infections post HSCT can also result in persistent cytopenias. Reactivation of human herpes virus 6 (HHV-6) and CMV in particular are associated with pancytopenia. HHV-6 reactivates at a median of 20 days post-HSCT and active infection has been shown in almost 50% of patients. The clinical syndrome associated with an active HHV-6 infection varies in intensity and may include encephalitis, rash, interstitial pneumonitis, and secondary graft failure. A transient, clinically insignificant HHV-6 reactivation occurs in many patients and because the symptoms of an HHV-6 infection are heterogenous and therefore less recognized, the disease may become severe prior to the recognition that the reactivation requires treatment. HHV-6 can become chronically active and has been associated not only with secondary graft failure, but pure red cell aplasia as well.

CMV reactivation in the post HSCT period can also be accompanied by an acute syndrome manifested by fever, myalgia, and suppressed marrow function. Leukopenia at the start of CMV therapy has been associated with a poor response to anti-viral therapy and is a risk factor for progression of CMV viremia to CMV disease. While the most serious manifestations of CMV disease are related to pulmonary and enteral infections CMV-induced marrow suppression and marrow failure has been described, with identification of specific genotypes of CMV highly associated with mortality from pancytopenia. Because CMV and the treatment for CMV can both be associated with post HSCT cytopenias, it is often difficult to distinguish which of the two is the major etiological factor.

Although the pathophysiology is unclear, persistent cytopenias post HSCT have also been associated with acute and chronic GVHD, bacterial and fungal infections, and impaired hepatic and renal function. Because failure of hematopoietic recovery after HSCT is associated with compromised patient survival, this protocol was developed to provide patients with persistent cytopenias post HSCT a boost of their original donors' HSCs to improve peripheral blood counts.

ELIGIBILITY:
Inclusion Criteria:

1. No evidence of active disease as measured by staging studies pertinent to the particular diagnosis within 1 month of the CD 34+ boost
2. Full donor chimerism as manifested by a ≥ 90% donor peripheral blood total, MNC, and T cell chimerism result on the last two studies prior to the planned CD 34+ boost, with the second study performed within 1 month of the infusion.
3. HHV-6 and CMV negative by PCR for at least 1 month prior to the CD 34+ boost as measured by at least 2 assays within the month timeframe
4. ANC of < 1000 10^6/L or maintenance of an ANC ≥ 1000 10^6/L only with white cell growth factor support
5. Requirement for red cell transfusion to maintain a hemoglobin of ≥ 9.0 g/dL
6. Requirement for red cell transfusion to avoid symptomatic anemia in patients with hemoglobin values of ≤ 11.0 g/dL
7. Requirement for platelet transfusion to maintain a platelet count of ≥ 20 10^9/L
8. Requirement for platelet transfusion to avoid bleeding in patients with platelet counts ≤ 50 109/L
9. No signs of active acute GVHD (excluding stages I-II skin GVHD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Etiologies of post HSCT cytopenias | Up to 8 weeks
  Will be collected and reported descriptively.
CD34+/kg and CD3+/kg cell doses in the infused CD 34+ selected boost products | Up to 8 weeks
  Will be collected and reported descriptively.
Effects of the CD 34+ selected boost on peripheral blood cell counts | Up to 8 weeks
  Will be collected and reported descriptively.
Incidence of GVHD related to the CD34+ selected boost | Up to 8 weeks
  Will be collected and reported descriptively.
Incidence of grade 3-5 infusion reactions, graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0 | Up to 8 weeks
  Will be descriptive.
Incidence of severe GVHD (grades 3-4), graded according to standard criteria | Up to 8 weeks
  Will be descriptive.

CONTACTS AND LOCATIONS:
Overall Officials: Dolores Grosso, DNP, CRNP, Principal Investigator — Thomas Jefferson University

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org